CLINICAL TRIAL: NCT06420466
Title: Dietary Intake Status and Time-Restricted Feeding on Cardiovascular Health Effects in the Overweight Population: A Study of Students at a Shenzhen University
Brief Title: Time-Restricted Feeding on Cardiovascular Health Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhengqi Qiu (Other)
Collaborators: The Seventh Affiliated Hospital of Sun Yat-sen University (Other); Shenzhen University (Other)
Responsible Party: Sponsor-Investigator, Zhengqi Qiu, Associate researcher, Macau University of Science and Technology Hospital
Organization: Macau University of Science and Technology Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY-2022-101-01
Record Dates: First submitted 2024-05-04; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Time Restricted Feeding; Cardiovascular Health; Body Composition; Blood Pressure; Young Adult
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-restricted Feeding group (Experimental): Controlling the eating time to 6 hours per day, but not being prescriptive about the quantity and content of dietary intake.
  Interventions: Behavioral: Time-restricted Feeding
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Time-restricted Feeding — Controlling the eating time to 6 hours per day, but not being prescriptive about the quantity and content of dietary intake.
  Arms: Time-restricted Feeding group

SUMMARY:
Study Design and Participants This intervention study was conducted as a randomized controlled trial (RCT) aimed at investigating the effects of time-restricted feeding (TRF) on cardiovascular health markers among overweight male university students in Shenzhen, China. The study recruited male university students aged between 18 and 24 years, with a Body Mass Index (BMI) ranging from 24 to less than 28. All participants were free from severe psychiatric illnesses, metabolic syndrome, diabetes, alcoholic fatty liver disease, hyperthyroidism, or hypothyroidism. Inclusion criteria required participants to be non-smokers, not currently on any diet pills, and have no history of cardiovascular or metabolic diseases.

Randomization and Intervention Fifty eligible participants were randomly assigned to either the intervention group (n=25) or the control group (n=25). The intervention group underwent a 6-hour daily TRF from noon to 6 P.M., while the control group did not participate in TRF but maintained their usual eating patterns. No restrictions were placed on the type or quantity of food consumed by participants in either group.

Data Collection and Measures Body Composition and Anthropometry: Measurements included body mass index, body fat percentage, muscle mass, hydration levels, protein content, and visceral fat, all assessed using a bioelectrical impedance analysis scale (Mi Body Composition Scale 2 by Huami Technology). Waist circumference was manually measured by experienced nurses using a tape measure.

Blood Pressure and Heart Rate: These vital signs were monitored using an arm cuff electronic blood pressure monitor (Panasonic EW3153), with the arm positioned at heart level to ensure accuracy. Measurements were taken after at least five minutes of seated rest.

Nutritional Intake Although time-restricted feeding interventions do not usually change the content or quantity of dietary intake, the total daily intakes of energy, fat, protein, carbohydrate, cholesterol, and fibre were calculated using the Nutritionist Pro food analysis program. This was used to determine possible changes in the subjects' dietary composition as a result of the intervention.

Compliance and Ethical Considerations The study protocol was approved by the Ethics Committee of the Seventh Affiliated Hospital of Sun Yat-sen University (Shenzhen), with the approval number KY-2022-101-01. All data were handled confidentially, and measures were taken to ensure high adherence and minimal loss to follow-up.

Statistical Analysis Descriptive statistics such as range, mean, standard deviation, and percentages were used to describe the sample characteristics. To compare differences, the change from baseline levels was assessed to account for initial variability, employing an independent samples t-test for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were able to provide signed and dated written informed consent.
* Subjects are male undergraduates aged 18-24 years old.
* BMI between 24 and 28.
* Normal sleep duration, usually between 7-9 hours per day.
* Stable sleep habits, typically going to bed around midnight (±1 hour).

Exclusion Criteria:

* Inability to comply with the time-limited diet plan.
* Experiencing hypoglycemic reactions during the time-limited diet program.
* Presence of metabolic diseases such as diabetes.
* Participation in high-intensity physical training for more than 5 hours per week.
* Extreme chronotypes, as indicated by scores ≤30 or ≥70 on the Morning and Evening Questionnaire Self-Assessment Scales (MEQ-SA).
* Severe weight instability, defined as weight gain or loss of more than 5 kg in the 3 months prior to the study.
* Severe food allergy or intolerance.
* Participation in another medical study within 6 months prior to the first study visit.

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — A single physiological group of others was chosen for the study because dietary habits and physiological indicators may differ between genders.
Enrollment: 50 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | 4 Weeks
  BMI is calculated using a standardized ratio of weight to height (kg/m²), offering a quantitative measure of body composition. This outcome will be assessed using digital scales for accurate weight measurement and stadiometers for height, ensuring precise BMI calculation.
Waist Circumference | 4 Weeks
  Waist circumference is measured using a flexible measuring tape, which allows for a direct quantification of visceral fat accumulation. This measure provides critical insights into metabolic health risks, differentiating it from BMI by focusing specifically on central obesity.
Blood pressure | 4 Weeks
  Revised Description: Blood pressure will be measured using a standardized sphygmomanometer, ensuring consistent and reproducible results. This tool will help monitor changes in systolic and diastolic blood pressure, which are vital for evaluating the effects of time-restricted eating on cardiovascular health.
Nutritional indicators | 4 Weeks
  Nutritional indicators will be assessed through detailed 24-hour dietary recall interviews and food diaries analyzed using nutritional analysis software. This approach will quantify changes in nutrient intake, highlighting the dietary impact of time-restricted feeding interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen university, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
No external funding was received for this study and there are no plans to make individual participant data available to other researchers